CLINICAL TRIAL: NCT01785459
Title: Treatment of Benign Headache in the Emergency Department Population With Lower Cervical Paraspinous Bupivacaine Injections Versus Anti-Emetic Treatment in the Emergency Department Population: Randomized Prospective Control Trial
Brief Title: Bupivacaine for Benign Headache in the ED
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to enroll adequate number of patients.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBH-001
Record Dates: First submitted 2013-02-03; First posted 2013-02-07 (Estimated); Results first posted 2019-04-03 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2019-03

CONDITIONS: Benign Headache
Keywords: headache; migraine; bupivacaine
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — Bupivacaine; Standard of Care; Prochlorperazine; Metoclopramide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard care (Active Comparator): intravenous Prochlorperazine
  Interventions: Drug: Standard Care
- treatment (Experimental): 0.5% bupivacaine
  Interventions: Drug: 0.5% bupivacaine

INTERVENTIONS:
Drug: 0.5% bupivacaine — The injection site will be prepared using common sterile technique with 2% chlorhexidine. 1.5 mL of 0.5% bupivacaine will be will be injected bilaterally in the paraspinal musculature of the cervical spine. Location would be approximately 1 cm superior to spinous process of C7 and approximately 2-3 cm laterally. The needle is inserted 1 to 1.5 inches into the paraspinous musculature at this level. A 27-gauge needle would be used to minimize tissue trauma and pain to the patient. Our method of injection is followed quite closely with the technique depicted in multiple retrospective studies. We chose to follow previous reported technique secondary to good clinical efficacy and impressive documented safety profile. Additionally, before injection, aspiration would be performed to lesson chance of intravascular injection.
  Arms: treatment
Drug: Standard Care — 10 mg Intravenous injection of Prochlorperazine
  Other Names: Prochlorperazine; Reglan
  Arms: standard care

SUMMARY:
Headache is a common chief complaint of patients presenting to the emergency department (ED), accounting for approximately 3 million ED visits per year. Headache treatment is often a source of frustration for both patients and providers. By the time patients with benign headaches arrive in the emergency department, they have often failed non-invasive therapeutic attempts and providers are often left with few therapeutic options. Treatment of benign headache varies between providers, often including systemic medications with a multitude of possible side effects. In recent years, there has been preliminary investigation into anesthetic injections for the undifferentiated headache patient presenting to the emergency department. It has been proposed that these patients presenting with benign headache might benefit from this novel treatment.

Patients that present to the Emergency Department with a diagnosis of benign or primary headache with serious or life-threatening causes of headache will be offered enrollment into the study.

Following consent, subjects will receive either 0.5% bupivacaine injected bilaterally in the paraspinal musculature of the cervical spine or the standard treatment with intravenous Prochlorperazine. The subjects will complete a validated pain scale before, and 20 minutes after injection. At twenty minutes post-injection, the subject will be reevaluated for symptoms. The subject will then be eligible for discharge or standard treatment at the discretion of the treating physician.

Subjects will be followed for 72 hours after enrollment for headache recurrence. Subjects will be monitored for immediate and post-discharge complications.

DETAILED DESCRIPTION:
Headache is a common chief complaint of patients presenting to the emergency department (ED), accounting for approximately 3 million ED visits per year. Headache treatment is often a source of frustration for both patients and providers. By the time patients with benign headaches arrive in the emergency department, they have often failed non-invasive therapeutic attempts and providers are often left with few therapeutic options. Treatment of benign headache varies between providers, often including systemic medications with a multitude of possible side effects. Additionally, most headache cocktails require prolonged duration of treatment, occupying valuable bed space in increasingly busy emergency departments.

In recent years, there has been preliminary investigation into anesthetic injections for the undifferentiated headache patient presenting to the emergency department. It has been proposed that these patients presenting with benign headache might benefit from this novel treatment. Since 2003, paraspinal muscle injections of bupivacaine have been used in emergency department patients with encouraging results. The mechanism of action is not clearly understood; however, it has been proposed that these injections affect the trigeminocervical complex hypothesized to play an integral role in headache physiology, similar to the same mechanism behind greater occipital nerve blocks used by neurologists.

To the best of the investigators knowledge, there has never been a prospective double-blinded randomized control trial addressing this novel approach to headache management. Even so, the topic of using bupivacaine to inject the paraspinal musculature of the cervical spine has gained wider recognition over the past year. The topic has been discussed heavily on emergency medicine blogs and podcasts. Additionally, online videos have been posted to educate emergency medicine providers on the injection technique. According to retrospective literature, clinical efficacy was observed with a significant proportion of the patients receiving therapeutic effect. These studies, along with anecdotal experience with the procedure at the investigators institution, have led to great excitement concerning the possibility of a new approach to emergency department headache management. However, the topic still needs investigation with a well-designed prospective clinical trial to determine true clinical utility.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old
2. Diagnosis of benign or primary headache

Exclusion Criteria:

1. Hypersensitivity or allergy to bupivacaine (amide anesthetics) or prochlorperazine or other drugs in the same class, dopaminergic blockers.
2. Overlying signs of infection at site of injection (Erythema, purulence, open skin)
3. Neck pathology ( History of surgery to the cervical spine, History of surgical hardware in place, Documented disc abnormality, History of vertebral artery or carotid artery dissection, Torticollis)
4. Intracranial abnormality/pathology (Tumor, Hemorrhage, Concussion or post concussive syndrome)
5. History of increased intracranial pressure (ICP)
6. A known history of extrapyramidal symptoms, dystonia, parkinsonism, tardive dyskinesia or neuroleptic malignant syndrome
7. Known pregnancy
8. Narcotic seeking patients as determined by the treating physician with optional assistance from medical record review and North Carolina Drug Database

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Fox, MD, Principal Investigator — Carolinas Medical Center; Carey Nichols, MD, Principal Investigator — Carolinas Medical Center
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Care | Treatment
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Treatment | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (10.5) | 30 (9.1) | 32 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 1 | 6 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 4 | 1 | 5
  African American | 6 | 10 | 16
  Hispanic | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Length of Stay
Description: Length of stay will be calculated as total time of encounter as well as time from doctor encounter to disposition decision
Time Frame: enrollment day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Standard Care | Treatment
Number analyzed (Participants) | 11 | 12
minutes | 158 (85.5) | 131 (113.5)

2. Primary Outcome: Incidence of Immediate and Post-discharge Complications.
Description: Subjects will be monitored for both immediate and post discharge complications up to 72 hours after enrollment that include: persistent local pain, bleeding, infection, and inadvertent intravascular injection resulting in seizure or possible cardiovascular collapse.
Time Frame: 72 hours
Population: See AE results
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Treatment
Number analyzed (Participants) | 11 | 12
Participants | 1 | 2

3. Secondary Outcome: Symptomatic Relief of Headache
Description: Symptomatic relief of headache will be measured by:
  1. Change from pre-intervention pain using a visual analog scale and ordinal scale:
     1. Headache relief
     2. Partial headache relief
     3. No headache relief
     4. Headache worsened
  2. Treatment failure, defined as requirement for additional medication administered in the ED due to incomplete pain relief from the paraspinous bupivacaine injections or the initial dose of intravenous prochlorperazine.
  3. Repeat visit for headache pain within 72 hour time period, excluding routine follow up care, determined by electronic medical record review and telephone follow up.
Time Frame: 20 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Treatment
Number analyzed (Participants) | 11 | 12
Participants
  Headache relief | 7 | 9
  Partial headache relief | 3 | 2
  No headache relief | 1 | 0
  Headache worsened | 0 | 1

ADVERSE EVENTS:
Time Frame: 72 hours and immediately following injection
Arm/Group | Standard Care | Treatment
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 1/11 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=11) | Treatment (N=12)
pain with injection (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Akathesia (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No